CLINICAL TRIAL: NCT00695669
Title: A Trial to Evaluate the Immunogenicity of Accelerated Primary Vaccination With Monovalent A/Indonesia/5/05 (H5N1) Vaccine Antigen in Association With AS03 Adjuvant in Adults Aged 18-64
Brief Title: A Trial to Test the Response to Different Vaccination Regimens With an H5N1 Vaccine With AS03 in Adults Aged 18-64
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111626
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: H5N1; immunogenicity; influenza; Avian; pandemic; vaccines; human; safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Influenza A (H5N1) 1 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine
- Influenza A (H5N1) 2 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, at Day 0 and Day 14. The vaccine was administered intramuscularly in the deltoid region of the arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine
- Influenza A (H5N1) 3 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, at Day 0 and Day 7. The vaccine was administered intramuscularly in the deltoid region of the arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine
- Influenza A (H5N1) 4 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, at Day 0. The vaccine was administered intramuscularly in the deltoid region of the arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus Monovalent Vaccine — Two doses administered intramuscularly (IM), the first in the deltoid region of the non-dominant arm and the second in the deltoid region of the dominant arm.

SUMMARY:
The purpose of the study is to characterize the immunogenicity & safety of 2 doses of GSK's avian flu vaccine GSK 1557484A given according to different regimens to adults aged 18 to 64 years

DETAILED DESCRIPTION:
A Phase 2, open-label, randomized, parallel group, multi-centered study designed to evaluate the immunogenicity and safety of a 2-dose series of avian influenza vaccine plus AS03 adjuvant according to different regimens, in adults aged 18-64 years. All subjects will receive active study vaccine; no subjects are to receive placebo. A total of 312 subjects will be enrolled in this study at approximately 3 study centers in Canada. All subjects will attend formal study center visits for safety and immunogenicity assessments on Days 0, 21, 42, and 182. Additional formal study center visits will be scheduled at additional timepoints for subjects in particular dose groups. In addition, a telephone call will be conducted for all subjects on Day 51

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18-64 years old at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Good general health as established by medical history and clinical examination before entering into the study.
* Access to a consistent means of telephone contact.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of short- and long-term safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study

Exclusion Criteria:

* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may be enrolled, but other histological types of skin cancer are exclusionary.
* Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may be enrolled.
* Presence of an oral temperature ≥37.8ºC, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 1 month of study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Administration of any vaccines within 30 days before study enrollment or during the 30 days following the last test article dose. Subjects who receive such immunizations on an emergent basis after enrollment will be followed per protocol and included in the Total Vaccinated Cohort (TVC), but excluded from the According to Protocol (ATP) Cohort for both safety and immunogenicity.
* Previous administration of any H5N1 vaccine.
* Use of any investigational or non-registered product (drug or vaccine) or planned participation in another investigational study within 30 days prior to study enrollment, or during the 182 days following the first test article dose. Use of any investigational or non-registered product with immunosuppressive properties is exclusionary at any time during the trial.
* Receipt of any immunoglobulins and/or any blood products within 6 months of study enrollment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins or mercurial preservatives); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result prior to either vaccination.
* Lactating or nursing.
* Women of child bearing potential who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to treatments. Note: all women will have urine pregnancy tests regardless of their status.
* Known receipt of analgesic or antipyretic medication on the day of treatment with specific intent of prophylaxis of vaccine reactogenicity on the day of first or any treatment. Subjects on stable chronic regimens of potentially analgesic or anti-pyretic medications for pre-existing diagnoses are not required to discontinue them

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2008-06-05; Primary Completion 2008-08-13 (Actual); Study Completion 2009-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Canada (3):
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lasko B, Reich D, Madan A, Roman F, Li P, Vaughn D. Rapid immunization against H5N1: a randomized trial evaluating homologous and cross-reactive immune responses to AS03(A)-adjuvanted vaccination in adults. J Infect Dis. 2011 Aug 15;204(4):574-81. doi: 10.1093/infdis/jir328. PMID 21791660
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111626 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Started | 78 | 78 | 78 | 78
Completed | 74 | 74 | 75 | 74
Not Completed | 4 | 4 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 4 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group | Total
Number analyzed (Participants) | 78 | 78 | 78 | 78 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (13.88) | 39.7 (13.81) | 40.8 (13.87) | 40.7 (13.22) | 40.3 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 43 | 48 | 166
  Male | 39 | 42 | 35 | 30 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination (Day 0) reciprocal hemagglutination inhibition (HI) titer less than (<) 1:10 and a post-vaccination (at Day 14 post Dose 2) reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal HI titer ≥ 1:10 and at least a four-fold increase in post-vaccination (at Day 14 post Dose 2) titer.
Time Frame: At Day 14 post Dose 2
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data for the primary outcome variables were available i.e. all subjects had to have at least Day 0 and post-vaccination HI titer results for the A/Indonesia/5/05 virus.
Measure: Number; unit: Subjects
Groups:
- Influenza A (H5N1) 3 Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted,at Day 0 and Day 7. The vaccine was administered intramuscularly in the deltoid region of the arm.
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 69 | 74 | 75
Subjects | 63 | 64 | 53 | 54

2. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The Confidence Interval for this outcome was 98.75%.
Time Frame: At Day 0 and at Day 14 post Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 69 | 74 | 75
titers
  H5N1 at Day 0 | 5.4 [4.7 to 6.1] | 5.3 [4.7 to 6.0] | 5.5 [4.8 to 6.3] | 5.8 [4.8 to 7.0]
  H5N1 at Day 14 post Dose 2 | 640.0 [413.7 to 990.0] | 345.0 [221.2 to 538.1] | 77.7 [49.9 to 121.0] | 67.4 [42.5 to 107.0]

3. Primary Outcome: Number of Seroprotected Subjects Against 3 Strains the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40.
Time Frame: At Day 0 and at Day 14 post Dose 2
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 69 | 74 | 75
Subjects
  H5N1 at Day 0 | 2 | 1 | 2 | 3
  H5N1 at Day 14 post Dose 2 | 63 | 64 | 55 | 56

4. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 1 Group.
Time Frame: At Days 0, 21, 28, 35, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 1 Group
Number analyzed (Participants) | 65
titers
  H5N1 at Day 0 [N=65] | 5.4 [4.9 to 5.9]
  H5N1 at Day 21 [N=64] | 40.2 [27.9 to 58.1]
  H5N1 at Day 28 [N=65] | 150.9 [101.1 to 225.1]
  H5N1 at Day 35 [N=65] | 640.0 [455.9 to 898.4]
  H5N1 at Day 42 [N=62] | 523.3 [366.0 to 748.3]
  H5N1 at Day 182 [N=65] | 51.1 [37.0 to 70.6]

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 2 Group.
Time Frame: At Days 0, 14, 21, 28, 35, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 2 Group
Number analyzed (Participants) | 69
titers
  H5N1 at Day 0 [N=69] | 5.3 [4.9 to 27.5]
  H5N1 at Day 14 [N=68] | 26.8 [18.8 to 38.0]
  H5N1 at Day 21 [N=69] | 99.8 [67.0 to 148.8]
  H5N1 at Day 28 [N=69] | 345.0 [244.2 to 487.5]
  H5N1 at Day 35 [N=69] | 305.9 [220.8 to 423.7]
  H5N1 at Day 42 [N=68] | 262.3 [192.9 to 356.8]
  H5N1 at Day 182 [N=68] | 36.5 [27.5 to 48.4]

6. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 3 Group.
Time Frame: At Days 0, 7, 14, 21, 28, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 3 Group
Number analyzed (Participants) | 74
titers
  H5N1 at Day 0 [N=74] | 5.5 [4.9 to 6.1]
  H5N1 at Day 7 [N=74] | 7.6 [6.1 to 9.4]
  H5N1 at Day 14 [N=73] | 45.1 [32.0 to 63.5]
  H5N1 at Day 21 [N=74] | 77.7 [55.1 to 109.7]
  H5N1 at Day 28 [N=72] | 99.8 [70.9 to 140.6]
  H5N1 at Day 42 [N=73] | 81.1 [58.7 to 112.0]
  H5N1 at Day 182 [N=71] | 21.3 [16.2 to 28.1]

7. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 4 Group.
Time Frame: At Days 0, 7, 14, 21, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 75
titers
  H5N1 at Day 0 [N=75] | 5.8 [5.0 to 6.7]
  H5N1 at Day 7 [N=74] | 10.8 [8.0 to 14.6]
  H5N1 at Day 14 [N=75] | 67.4 [47.1 to 96.6]
  H5N1 at Day 21 [N=74] | 76.3 [52.6 to 110.8]
  H5N1 at Day 42 [N=74] | 78.9 [55.8 to 111.5]
  H5N1 at Day 182 [N=73] | 28.2 [21.0 to 37.8]

8. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 1 Group.
Time Frame: At Days 0, 21, 28, 35, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 1 Group
Number analyzed (Participants) | 65
titers
  VIET at Day 0 [N=65] | 5.3 [4.9 to 5.8]
  VIET at Day 21 [N=64] | 9.7 [7.3 to 12.9]
  VIET at Day 28 [N=65] | 20.7 [15.0 to 28.6]
  VIET at Day 35 [N=65] | 61.6 [44.4 to 85.6]
  VIET at Day 42 [N=62] | 48.6 [34.7 to 68.1]
  TURK at Day 0 [N=65] | 7.6 [6.0 to 9.7]
  TURK at Day 21 [N=64] | 22.5 [16.5 to 30.8]
  TURK at Day 28 [N=65] | 46.4 [32.0 to 67.4]
  TURK at Day 35 [N=65] | 181.8 [131.9 to 250.7]
  TURK at Day 42 [N=62] | 162.7 [120.9 to 218.9]
  TURK at 182 [N=65] | 25.8 [19.1 to 35.0]

9. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 2 Group.
Time Frame: At Days 0, 14, 21, 28, 35, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 2 Group
Number analyzed (Participants) | 69
titers
  VIET at Day 0 [N=69] | 5.4 [5.0 to 5.9]
  VIET at Day 14 [N=68] | 9.2 [7.2 to 11.7]
  VIET at Day 21 [N=69] | 15.1 [11.2 to 20.3]
  VIET at Day 28 [N=69] | 29.9 [21.8 to 40.9]
  VIET at Day 35 [N=69] | 26.5 [19.9 to 35.2]
  VIET at Day 42 [N=68] | 23.2 [17.4 to 30.9]
  TURK at Day 0 [N=69] | 7.1 [5.7 to 8.9]
  TURK at Day 14 [N=68] | 17.0 [12.0 to 24.0]
  TURK at Day 21 [N=69] | 36.4 [25.4 to 52.1]
  TURK at Day 28 [N=69] | 83.7 [59.2 to 118.4]
  TURK at Day 35 [N=69] | 74.9 [54.7 to 102.5]
  TURK at Day 42 [N=68] | 68.3 [50.5 to 92.4]
  TURK at Day 182 [N=68] | 18.5 [14.1 to 24.4]

10. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 3 Group.
Time Frame: At Days 0, 7, 14, 21, 28, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 3 Group
Number analyzed (Participants) | 74
titers
  VIET at Day 0 [N=74] | 5.3 [4.9 to 5.8]
  VIET at Day 7 [N=74] | 6.4 [5.6 to 7.4]
  VIET at Day 14 [N=73] | 13.7 [10.4 to 17.9]
  VIET at Day 21 [N=74] | 16.1 [12.2 to 21.2]
  VIET at Day 28 [N=72] | 15.3 [11.6 to 20.1]
  VIET at Day 42 [N=73] | 13.4 [10.5 to 17.1]
  TURK at Day 0 [N=74] | 7.2 [5.9 to 8.9]
  TURK at Day 7 [N=74] | 8.7 [6.8 to 11.2]
  TURK at Day 14 [N=73] | 27.2 [19.9 to 37.3]
  TURK at Day 21 [N=74] | 33.5 [23.9 to 46.7]
  TURK at Day 28 [N=72] | 34.9 [25.2 to 48.4]
  TURK at Day 42 [N=73] | 34.7 [24.9 to 48.4]
  TURK at Day 182 [N=71] | 13.7 [10.6 to 17.7]

11. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 4 Group.
Time Frame: At Days 0, 7, 14, 21, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 75
titers
  VIET at Day 0 [N=75] | 5.8 [5.1 to 6.6]
  VIET at Day 7 [N=74] | 7.9 [6.4 to 9.8]
  VIET at Day 14 [N=75] | 16.3 [12.1 to 21.9]
  VIET at Day 21 [N=74] | 16.2 [12.1 to 21.6]
  VIET at Day 42 [N=74] | 16.0 [12.3 to 20.6]
  TURK at Day 0 [N=75] | 7.7 [6.2 to 9.4]
  TURK at Day 7 [N=74] | 11.8 [8.7 to 16.0]
  TURK at Day 14 [N=75] | 28.9 [20.5 to 40.8]
  TURK at Day 21 [N=74] | 31.2 [22.4 to 43.5]
  TURK at Day 42 [N=74] | 35.6 [25.9 to 48.9]
  TURK at Day 182 [N=73] | 16.4 [12.4 to 21.7]

12. Secondary Outcome: Number of Seroconverted Subjects Against the A/Indonesia/5/2005 (H5N1), Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination (Day 0) reciprocal HI titer < 1:10 and a post-vaccination (at Day 14 post Dose 2) reciprocal titer ≥ 1:40 or a pre-vaccination reciprocal HI titer ≥ 1:10 and at least a four-fold increase in post-vaccination (at Day 14 post Dose 2) titer.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 62 | 78 | 73 | 74
Subjects
  H5N1 | 59 | 63 | 57 | 55
  VIET | 41 | 35 | 16 | 19
  TURK | 52 | 51 | 41 | 39

13. Secondary Outcome: Number of Seroconverted Subjects Against the A/Indonesia/5/2005 (H5N1) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination (Day 0) reciprocal hemagglutination inhibition (HI) titer < 1:10 and a post-vaccination (at Day 14 post Dose 2) reciprocal titer ≥ 1:40 or a pre-vaccination reciprocal HI titer ≥ 1:10 and at least a four-fold increase in post-vaccination (at Day 14 post Dose 2) titer.
Time Frame: At Day 182
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 68 | 71 | 73
Subjects
  H5N1 | 45 | 42 | 29 | 38
  TURK | 30 | 22 | 14 | 18

14. Secondary Outcome: Geometric Mean Fold-rise (GMFR) for the A/Indonesia/5/2005 (H5N1), Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: The GMFR is presented as the GMT ratio between GMTs at Day 42/182 and at Day 0.
Time Frame: At Days 0, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 68 | 73 | 74
Fold increase
  H5N1 at Day 42 [N=62,68,73,74] | 97.3 [67.1 to 141.2] | 49.4 [36.0 to 67.7] | 14.8 [10.6 to 20.5] | 13.5 [9.4 to 19.4]
  H5N1 at Day 182 [N=65,68,71,73] | 9.5 [6.9 to 13.2] | 6.9 [5.2 to 9.1] | 3.9 [2.9 to 5.1] | 4.8 [3.6 to 6.5]
  VIET at Day 42 [N=62,68,73,74] | 9.1 [6.5 to 12.8] | 4.3 [3.2 to 5.7] | 2.5 [2.0 to 3.2] | 2.7 [2.2 to 3.5]
  TURK at Day 42 [N=62,68,73,74] | 21.7 [15.1 to 31.3] | 9.6 [6.8 to 13.4] | 4.8 [3.4 to 6.6] | 4.6 [3.4 to 6.3]
  TURK at Day 182 [N=65,68,71,73] | 3.4 [2.5 to 4.6] | 2.7 [2.0 to 3.7] | 1.9 [1.5 to 2.6] | 2.1 [1.6 to 2.8]

15. Secondary Outcome: Micro-neutralization (MN) Titers for Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 1 Group.
Time Frame: At Days 0, 21, 28, 35, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 1 Group
Number analyzed (Participants) | 65
titers
  VIET at Day 0 [N=65] | 31.8 [24.3 to 41.4]
  VIET at Day 21 [N=64] | 85.0 [65.0 to 111.1]
  VIET at Day 28 [N=65] | 99.8 [78.2 to 127.3]
  VIET at Day 35 [N=65] | 142.6 [113.7 to 178.8]
  VIET at Day 42 [N=62] | 151.3 [120.3 to 190.3]
  TURK at Day 0 [N=65] | 26.5 [20.1 to 35.1]
  TURK at Day 21 [N=64] | 57.5 [43.7 to 75.6]
  TURK at Day 28 [N=65] | 139.9 [102.5 to 191.1]
  TURK at Day 35 [N=65] | 442.6 [343.6 to 570.3]
  TURK at Day 42 [N=62] | 377.0 [296.1 to 480.0]
  TURK at Day 182 [N=65] | 245.5 [186.2 to 323.5]

16. Secondary Outcome: Micro-neutralization (MN) Titers for Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 2 Group.
Time Frame: At Days 0, 14, 21, 28, 35, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 2 Group
Number analyzed (Participants) | 69
titers
  VIET at Day 0 [N=69] | 34.5 [27.7 to 42.8]
  VIET at Day 14 [N=69] | 99.4 [80.6 to 122.5]
  VIET at Day 21 [N=69] | 104.3 [85.4 to 127.4]
  VIET at Day 28 [N=69] | 146.9 [119.6 to 180.4]
  VIET at Day 35 [N=69] | 142.0 [119.1 to 169.4]
  VIET at Day 42 [N=68] | 134.5 [109.0 to 166.0]
  TURK at Day 0 [N=69] | 24.1 [20.0 to 29.1]
  TURK at Day 14 [N=68] | 64.9 [49.6 to 84.9]
  TURK at Day 21 [N=69] | 107.0 [82.0 to 139.7]
  TURK at Day 28 [N=69] | 224.0 [183.4 to 273.4]
  TURK at Day 35 [N=69] | 221.7 [181.9 to 270.3]
  TURK at Day 42 [N=68] | 227.8 [187.0 to 277.6]
  TURK at Day 182 [N=68] | 230.2 [184.2 to 287.6]

17. Secondary Outcome: Micro-neutralization (MN) Titers for Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 3 Group.
Time Frame: At Days 0, 7, 14, 21, 28, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 3 Group
Number analyzed (Participants) | 74
titers
  VIET at Day 0 [N=74] | 32.9 [26.0 to 41.6]
  VIET at Day 7 [N=74] | 42.2 [33.5 to 53.1]
  VIET at Day 14 [N=73] | 125.5 [96.4 to 163.3]
  VIET at Day 21 [N=74] | 133.8 [103.1 to 173.8]
  VIET at Day 28 [N=72] | 119.4 [93.6 to 152.3]
  VIET at Day 42 [N=73] | 114.5 [91.2 to 143.7]
  TURK at Day 0 [N=74] | 23.4 [18.7 to 29.4]
  TURK at Day 7 [N=74] | 25.1 [20.3 to 31.1]
  TURK at Day 14 [N=73] | 83.6 [61.6 to 113.5]
  TURK at Day 21 [N=74] | 105.8 [80.0 to 140.0]
  TURK at Day 28 [N=72] | 115.5 [87.0 to 153.4]
  TURK at Day 42 [N=73] | 146.7 [118.3 to 182.0]
  TURK at Day 182 [N=71] | 138.7 [105.9 to 181.8]

18. Secondary Outcome: Micro-neutralization (MN) Titers for Antibodies Against the Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). This outcome only covers results for the Pumarix 4 Group.
Time Frame: At Days 0, 7, 14, 21, 42 and 182.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 75
titers
  VIET at Day 0 [N=75] | 36.1 [28.4 to 45.8]
  VIET at Day 7 [N=74] | 62.8 [48.3 to 81.5]
  VIET at Day 14 [N=75] | 135.6 [106.9 to 171.9]
  VIET at Day 21 [N=74] | 109.3 [85.3 to 140.0]
  VIET at Day 42 [N=74] | 93.7 [72.3 to 121.4]
  TURK at Day 0 [N=75] | 24.3 [19.6 to 30.1]
  TURK at Day 7 [N=74] | 36.5 [27.8 to 47.8]
  TURK at Day 14 [N=75] | 97.2 [74.2 to 127.3]
  TURK at Day 21 [N=74] | 97.5 [75.3 to 126.4]
  TURK at Day 42 [N=74] | 132.1 [103.1 to 169.3]
  TURK at Day 182 [N=73] | 147.3 [112.9 to 192.3]

19. Secondary Outcome: Number of Subjects With a Vaccine Response of MN Assessed Antibodies for Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: Subjects with a vaccine response were defined as vaccinated subjects who had either a pre-vaccination titer < 1:28 and a post vaccination titer ≥ 1:56 or a pre-vaccination titer ≥ 1:28 and at least a four-fold increase in post-vaccination titer.
Time Frame: At 7, 14 and 21 days after the second dose
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 69 | 74 | 75
Subjects
  VIET at 7 days post dose 2 [N=65,69,72,74] | 28 | 26 | 34 | 16
  VIET at 14 days post dose 2 [N=65,69,73,75] | 35 | 36 | 33 | 32
  VIET at 21 days post dose 2 [N=62,69,71,74] | 33 | 32 | 33 | 33
  TURK at 7 days post dose 2 [N=65,69,73,74] | 37 | 37 | 33 | 11
  TURK at 14 days post dose 2 [N=65,69,74,75] | 54 | 54 | 43 | 35
  TURK at 21 days post dose 2 [N=62,69,72,74] | 50 | 53 | 40 | 37

20. Secondary Outcome: Number of Subjects With a Vaccine Response of MN Assessed Antibodies for Flu A/Vietnam/1194/2004 (VIET) and Flu A/Turkey/Turkey/1/2005 (TURK) Strains of Influenza Disease.
Description: as for outcome 19
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 62 | 68 | 73 | 74
Subjects
  VIET [N=62,68,72,74] | 33 | 34 | 30 | 24
  TURK [N=62,68,73,74] | 50 | 55 | 49 | 44

21. Secondary Outcome: Number of Subjects With a Vaccine Response of MN Assessed Antibodies for the Flu A/Turkey/Turkey/1/2005 (TURK) Strain of Influenza Disease.
Description: Subjects with vaccine response were defined as vaccinated subjects who had either a pre-vaccination titer < 1:28 and a post vaccination titer ≥ 1:56 or a pre-vaccination titer ≥ 1:28 and at least a four-fold increase in post-vaccination titer.
Time Frame: At Day 182
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 65 | 68 | 71 | 73
Subjects | 47 | 51 | 45 | 43

22. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any solicited local symptoms regardless of their intensity grade.
Time Frame: Within the 7-day follow-up period (Days 0-6) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one dose of vaccine and for whom any post-vaccination data were available and had the symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 76 | 77 | 78 | 77
Subjects
  Any Pain | 60 | 64 | 65 | 65
  Any Redness | 2 | 5 | 5 | 4
  Any Swelling | 4 | 5 | 5 | 3

23. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location (joint pain), muscle aches, shivering, sweating and fever. Fever was defined as oral temperature ≥ 38 degrees Celsius (°C). Any = occurrence of any solicited general symptoms regardless of intensity grade or relationship to vaccination.
Time Frame: Within the 7-day follow-up period (Days 0-6) after any vaccination
Population: as for outcome 22
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 76 | 77 | 78 | 77
Subjects
  Any Fatigue | 23 | 30 | 22 | 27
  Any Headache | 30 | 28 | 24 | 20
  Any Joint Pain | 20 | 23 | 22 | 11
  Any Muscle Aches | 49 | 43 | 40 | 40
  Any Shivering | 10 | 13 | 13 | 10
  Any Sweating | 15 | 11 | 8 | 5
  Any Fever | 2 | 4 | 1 | 1

24. Secondary Outcome: Number of Subjects With Medically Attended Adverse Events (MAEs).
Description: A MAE was defined as any unsolicited symptom that received medical attention such as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason.
Time Frame: From Day 0 to 182
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one dose of vaccine and for whom any post-vaccination data were available.
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Subjects | 18 | 19 | 15 | 21

25. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 51-day follow-up period (Days 0-50) after first vaccination.
Population: as for outcome 24
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Subjects | 34 | 37 | 41 | 27

26. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or resulted in a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to 182
Population: as for outcome 24
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Number analyzed (Participants) | 78 | 78 | 78 | 78
Subjects | 1 | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: Within the 7-day period after primary vaccination. Unsolicited AEs: Within the 51-day period after primary vaccination. SAEs: from Day 0 to Day 182.
Description: For solicited and general symptoms, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Influenza A (H5N1) 1 Group | Influenza A (H5N1) 2 Group | Influenza A (H5N1) 3 Group | Influenza A (H5N1) 4 Group
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/78 | 3/78 | 1/78
Other Adverse Events (participants affected / at risk) | 66/78 | 67/78 | 68/78 | 67/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza A (H5N1) 1 Group (N=78) | Influenza A (H5N1) 2 Group (N=78) | Influenza A (H5N1) 3 Group (N=78) | Influenza A (H5N1) 4 Group (N=78)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Influenza A (H5N1) 1 Group (N=78) | Influenza A (H5N1) 2 Group (N=78) | Influenza A (H5N1) 3 Group (N=78) | Influenza A (H5N1) 4 Group (N=78)
Pain (General disorders) | 60/76 | 64/77 | 65 | 65/77
Redness (General disorders) | 2/76 | 5/77 | 5 | 4/77
Swelling (General disorders) | 4/76 | 5/77 | 6 | 3/77
Fatigue (General disorders) | 23/76 | 30/77 | 22 | 27/77
Headache (General disorders) | 30/76 | 28/77 | 24 | 20/77
Joint pain (General disorders) | 20/76 | 23/77 | 22 | 11/77
Muscle aches (General disorders) | 49/76 | 43/77 | 40 | 40/77
Shivering (General disorders) | 10/76 | 13/77 | 13 | 10/77
Sweating (General disorders) | 15/76 | 11/77 | 8 | 5/77
Fever (General disorders) | 2/76 | 4/77 | 1 | 1/77
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 5 | 4 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 5 | 4
Nausea (Gastrointestinal disorders) | 1 | 5 | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 4 | 0
Injection site warmth (General disorders) | 2 | 0 | 1 | 4
Oedema peripheral (General disorders) | 0 | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.